CLINICAL TRIAL: NCT06914999
Title: Assessment of Radiation-Induced Vascular Complications in Patients With Head and Neck Cancers With PET/CT Imaging
Brief Title: Comparing an Investigational Scan (F-18 NaF PET/CT) to Standard of Care Imaging (F-18 FDG PET/CT) for Evaluating Vascular Complications in Patients Receiving Radiation Therapy for Head and Neck Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Amol Takalkar, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUDY00008261; NCI-2025-00404 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00008261 (Other: Emory University Hospital/Winship Cancer Institute); H-N Ca Patients (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2025-04-01; First posted 2025-04-07 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Head and Neck Squamous Cell Carcinoma; Hypopharyngeal Squamous Cell Carcinoma; Laryngeal Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Hypopharyngeal Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Hypopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Carcinoma | interventions — Fluorodeoxyglucose F18; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: For the purposes of this study, will contour the ascending aorta, arch of the aorta, carotid arteries, and descending aorta but these structures will not be a part of the treatment planning process and will be blinded to the treating physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (F-18 NaF PET/CT) (Experimental): Patients receive F-18 NaF IV and undergo PET/CT within 28 days of each SOC F-18 FDG PET/CT on study, once prior to initiation of SOC IMRT and once 12 weeks after completion of SOC IMRT.
  Interventions: Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Positron Emission Tomography; Drug: Sodium Fluoride F-18
- Arm II (F-18 NaF PET/CT) (Experimental): Patients receive F-18 NaF IV and undergo PET/CT within 28 days of each SOC F-18 FDG PET/CT on study, once prior to initiation of SOC IMPT and once 12 weeks after completion of SOC IMPT.
  Interventions: Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Intensity-Modulated Proton Therapy; Procedure: Positron Emission Tomography; Drug: Sodium Fluoride F-18

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Fludeoxyglucose F-18 — Given F-18 FDG
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Intensity-Modulated Proton Therapy — Undergo IMPT
  Other Names: IMPT
  Arms: Arm II (F-18 NaF PET/CT)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm I (F-18 NaF PET/CT)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Sodium Fluoride F-18 — Given IV
  Other Names: 18 F-NaF; F-18 NaF; Fluorine F 18 Sodium Fluoride; NaF F18; Sodium Fluoride F18

SUMMARY:
This early phase I trial compares sodium fluoride F-18 (F-18 NaF) positron emission tomography (PET)/computed tomography (CT) to the standard of care imaging scan (and fludeoxyglucose F-18 [F-18 FDG] PET/CT) for assessing the effects radiation therapy has on the blood vessels in the neck in patients with head and neck cancers. For people with cancers in the head and neck, doctors often use radiation to target both the tumor and nearby glands. Radiation therapy to this region can affect the blood vessels in the neck that supply blood to the brain. F-18 NaF and F-18 FDG are contrast agents that can be used together with PET/CT imaging to visualize areas inside the body. A PET scan is a procedure in which a small amount of radioactive glucose (sugar) is injected into a vein, and a scanner is used to make detailed, computerized pictures of areas inside the body where the glucose is taken up. A CT scan is a procedure that uses a computer linked to an x-ray machine to make a series of detailed pictures of areas inside the body. The pictures are taken from different angles and are used to create 3-dimensional views of tissues and organs. Combining a PET scan with a CT scan can help make the image easier to interpret. PET/CT scans are hybrid scanners that combine both modalities into a single scan during the same examination. Imaging with F-18 NaF PET/CT may be as effective or more effective than the standard F-18 FDG PET/CT for assessing the effects radiation therapy has on blood vessels in the neck in patients with head and neck cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the role of FDG- and NaF-PET in assessing radiation-induced vascular complications by comparing baseline and follow-up scans in patients with head and neck cancer.

II. To assess the presence and extent of radiation-induced vascular inflammation following proton versus (vs) photon radiation therapy (RT) in patients with head and neck cancer.

III. To determine the correlation between inflammation and actual radiation dose received to the vasculature to assess the effects of dose response.

SECONDARY OBJECTIVE:

I. To determine the effect of radiation-induced vascular inflammation (possibly atherosclerosis) on global brain function as measured by FDG-PET.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients receive F-18 NaF intravenously (IV) and undergo PET/CT within 28 days of each standard of care (SOC) F-18 FDG PET/CT on study, once prior to initiation of SOC intensity-modulated radiation therapy (IMRT) and once 12 weeks after completion of SOC IMRT.

ARM II: Patients receive F-18 NaF IV and undergo PET/CT within 28 days of each SOC F-18 FDG PET/CT on study, once prior to initiation of SOC intensity-modulated proton therapy (IMPT) and once 12 weeks after completion of SOC IMPT.

After completion of study intervention, patients are followed up within one to five business days.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age and older
* Diagnosis of clinical stage III-IVb (American Joint Committee on Cancer [AJCC] 8th edition) squamous cell carcinoma of the oropharynx (human papillomavirus [HPV]-negative), larynx, or hypopharynx, or clinical stage I-III (AJCC 8th edition) HPV-associated squamous cell carcinoma of the oropharynx receiving curative-intent, organ preservation (non-surgical)
* Treatment with concurrent chemoradiotherapy per institutional standard of care at the discretion of Medical Oncology. RT is delivered per institutional standard of care at the discretion of Radiation Oncology
* Patients must give protocol-specific consent on an Institutional Review Board (IRB)-approved consent form prior to completion of protocol-specific testing/procedures
* Women are eligible to participate in the study if they meet one of the following criteria:

  * Females of childbearing potential (FCBP) must have a negative pregnancy test at baseline and follow-up visit. Women of childbearing potential must undergo pregnancy testing during each study visit and agree to use at least one of the following methods of contraception throughout the study duration:

    * Oral contraceptives, transdermal contraceptives, injectable or implantable methods, intrauterine devices, and/or vaginal ring
    * Women who are postmenopausal (for at least one year), sterile, or hysterectomized;
    * Women who have undergone tubal ligation will be required to undergo pregnancy testing during each study visit

Exclusion Criteria:

* Adults who are unable to consent
* Pregnant women
* Prisoners
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier (i.e., have residual toxicities > grade 1)
* Patients who are receiving any other investigational agents or an investigational device within 21 days before administration of the F-18 NaF for the pre-RT PET/CT imaging
* Patients planned to receive any immunotherapy agent during their radiotherapy or in the interval between radiotherapy and post-RT PET/CT imaging
* History of allergic reactions attributed to compounds of similar chemical or biological composition to F-18 NaF or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Significant cardiovascular disease (eg, myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 3 months prior to study entry; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association class 3 or 4 congestive heart failure; or uncontrolled grade >= 3 hypertension (diastolic blood pressure >= 100 mmHg or systolic blood pressure >= 160 mmHg) despite antihypertensive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Radiation-induced vascular complications | Prior to and after undergoing radiation therapy, up to 6 months
  Will compare the presence and extent of radiation therapy (RT)-induced vascular complications between the two treatment modalities. The average standardized uptake volume (SUV) max and mean of fludeoxyglucose F-18 (FDG)- and sodium fluoride F-18 (NaF)-positron emission tomography (PET)/computed tomography (CT) scans pre- and post RT will be computed. Will assess the change in average SUVmax and SUVmean of FDG- and NaF-PET/CT scans pre- and post-RT. Will also assess the difference in average SUV mean between proton and photon RT. Will assess the difference in change in SUV mean between intensity-modulated radiation therapy (IMRT) and intensity-modulated photon therapy (IMPT) using a two-sample independent t-test or the Wilcoxon rank sum test for each SUVmean/max. A multivariable linear regression model with a backward elimination approach will be used to test the effect of clinicopathological variables on the change in SUVmax.
Radiation-induced vascular inflammation following IMRT or IMPT | Baseline up to 6 months
  Will evaluate the presence and extent of radiation-induced vascular inflammation following IMRT versus IMPT. Will determine the correlation between the actual radiation dose and radiation-induced vascular inflammation, measured by the average SUVmax/mean, and will be done using Pearson's correlation or Spearman's correlation analysis, as appropriate.
Percentage volumetric dose | Baseline up to 6 months
  The percentage volumetric dose will be recorded to determine the correlation between the actual radiation dose and the radiation-induced vascular inflammation, measured by the average SUVmax/mean, and will be done using Pearson's correlation or Spearman's correlation analysis, as appropriate.

SECONDARY OUTCOMES:
Total brain FDG uptake | Baseline up to 6 months
  Will assess the association of total brain FDG uptake between the two scanning methods (FDG and NaF PET/CT). The total brain FDG uptake pre- and post-RT will be measured. Will assess the association between the average SUVmax/mean difference of FDG- and NaF-PET/CT scans and the total brain FDG uptake. Will be performed using Pearson's correlation or Spearman's correlation analysis, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Amol M Takalkar, MD, MS, MBA, FACNM, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States